CLINICAL TRIAL: NCT06675110
Title: Diagnostic Tools for the Direct Detection of Orientia Tsutsugamushi
Brief Title: QuEST - Quick and Easy Scrub Typhus Diagnostic Tools
Acronym: QuEST
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OxTREC Reference: 4 - 24
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-01

CONDITIONS: Scrub Typhus
Keywords: Scrub typhus; Orientia tsutsugamushi; insulated isothermal PCR; diagnostic evaluation
MeSH Terms: conditions — Scrub Typhus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood in EDTA and clotted blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suscpected scrub typhus cases: Participants with symptoms and epidemiologic risks for of scrub typhus and testing positive by:
  1. StandardQ rapid diagnostic test OR
  2. InBios Scrub Typhus Detect IgM
  3. Insulated isothermal PCR

SUMMARY:
Evaluate the performance of insulated isothermal polymerase chain reaction (iiPCR) in the diagnosis of scrub typhus in Chiang Rai Province

DETAILED DESCRIPTION:
Screening and enrolment

The study team will screen patients presenting with fever at the out- and inpatient departments of study sites. A scrub typhus rapid diagnostic test (RDT) will be performed at all sites (e.g. Scrub Typhus IgM RDT, InBios International; Scrub Typhus IgM/IgA/IgG RDT, SDBioline; STANDARD Q Tsutsugamushi IgM/IgG, SDBiosensor) and insulated isothermal polymerase chain reaction (iiPCR) will be performed at Chiang Rai Clinical Research Unit (CCRU) central laboratories. Before being screened with any of the above tests for study purposes, potential participants will be asked to pre-consent to the screening test.

If participants have a positive screening test following an order form the treating physician as part of standard management (not for study purposes), this will be considered equivalent to a positive screening test; those subjects will be asked then to provide informed consent to participate in the study.

Eligible patients who agree to participate and/or their legal guardians will take part in the informed consent procedure. If the RDT or iiPCR test is positive for scrub typhus (one positive test is sufficient) or the patient has a fever and an eschar, the patient is formally enrolled into the study.

Every screened patient will receive a screening number and details are recorded into a screening log. Screening rejection is defined as patients who have been screened but are not enrolled into the study. Reasons for rejection may include any exclusion criteria, non-conformity with the inclusion criteria, or failure to obtain informed consent. Reasons will be recorded in the screening log. Patients who do not progress from screening to trial recruitment will not be assigned with a study number or have clinical data recorded in the screening log.

Inpatient stay Clinical review: Study patients will have their vital signs measured and recorded every 6 hours during hospitalisation. Details of antibiotics administered will be collected. Additional diagnostic test results (e.g. laboratory or imaging) requested by the medical team will also be collected and recorded on the case report from (CRF).

Patients admitted with scrub typhus to hospital for treatment will be discharged by the treating physician according to clinical improvement and resolution of fever.

Follow-up

Scheduled follow-up: A follow-up visits will occur at 2 weeks (+ 2 weeks). Examinations and samples are collected as outlined in the study flowchart (paragraph 3.3).

If the patient cannot be followed-up, then the reason for loss-to-follow-up will be recorded on the CRF.

Study participants are asked to contact the study team if fever and/or symptoms and signs compatible with scrub typhus appear after hospital discharge until the patient exits the study (after the 2 week follow-up appointment). Clinical findings and samples are collected as outlined in the study flowchart.

If the patient was discharged or leaves the hospital prior to cessation of fever, the patient will be given a tympanic membrane monitor and asked to measure their temperature 4 times a day (flexible/pragmatic timings) and record the results in a diary until their fever has cleared. The diary and the thermometer will be collected by the study team at follow-up and the temperature readings used to calculate the fever clearance time.

The performance of RDTs and of iiPCR will be compared to that of reference quantitative PCR (qPCR) and indirect immunofluorescence assay (IFA) for the diagnosis of scrub typhus on acute and paired (acute and convalescent) samples. The test will also be compared to the modified scrub typhus infection criteria (Paris et al., 2011)

ELIGIBILITY:
Inclusion Criteria:

* Acute (duration ≤14 days) fever (37.5°C or higher or a history of fever in the previous 24h) AND
* Eschar OR
* ≥ 2 of the following:
* Living in rural parts of Chiangrai Province or other ST risk areas
* History of outdoor risk activities in the 2 weeks before symptom onset
* Presenting during the rainy season or early cold season
* Two or more of: headache; myalgia, cough, abdominal symptoms (abdominal pain/ nausea-vomiting); myalgia; lymphadenopathy AND
* ≥ 7 years old AND
* Weight>15Kg AND
* The patient and/or where relevant their parent/guardian/caretaker/legally acceptable representative willing and able to give informed consent /assent for participation in the study AND Positivity to any of the screening tests (Immunochromatographic RDT or iiPCR)

Exclusion Criteria:

- Other clear focus of infection (e.g. lobar pneumonia by chest x-ray, abscess) OR Other clear cause of fever (e.g. positive Dengue IgM or NS1 antigen, positive blood cultures, untreated HIV)

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Febrile patients suspected of having scrub typhus and presenting to Mae Chan or Mae Suai district hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive- and negative predictive values of insulated isothermal polymerase chain reaction (iiPCR) compared to reference diagnostic tests | Baseline and week two

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Perrone, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Mae Chan District Hospital, Mae Chan, Changwat Chiang Rai, Thailand

IPD SHARING:
Plan to Share IPD: Yes
After publication of main findings, or 1 year after study completion (whichever comes first) and reasonable request to MORU data access committee